CLINICAL TRIAL: NCT02131766
Title: Unified Safety System (USS) Virginia Closed-Loop Versus Sensor Augmented Pump Therapy for Overnight Control in Type 1 Diabetes
Brief Title: USS Virginia Closed-Loop for Overnight Control in Type 1 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Sue Brown, Principal Investigator, University of Virginia
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 17351; 1DP3DK101055-01 (NIH); NCT02008188 (obsolete NCT alias)
Record Dates: First submitted 2014-05-02; First posted 2014-05-06 (Estimated); Results first posted 2020-04-16 (Actual); Last update posted 2020-04-16 (Actual); Status verified 2020-03

CONDITIONS: Diabetes Mellitus
Keywords: Diabetes Mellitus, Type 1; Artificial Pancreas Project (APP); Diabetes Assistant (DiAs); Closed-Loop Control (CLC)
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- USS Virginia Closed Loop Control (Experimental): The subject will be admitted to the research house/hotel and will be discharged after 5 nights. The subject will be trained on DiAs and on how to respond to the system's alerts. The DiAs will be initiated by 11:00 PM and will be discontinued before breakfast. The staff will be monitoring the subject remotely. The subject will need to remain within a 30 miles of the research house/hotel during the day and return by 6:00 PM.
  A limited number of UVA and UPadova subjects will be asked to wear the DiAs at home for 5 days at the conclusion of research house admission.
  Interventions: Device: DiAs
- Sensor Augmented Pump Therapy (Placebo Comparator): The subject will wear the continuous glucose monitor with the study insulin pump for a full 7 day period (approximately 7 consecutive 24 hour periods). The subject will follow their usual regimen. The subject will be asked to use the bolus calculator function on your insulin pump and enter the carbohydrate information that you eat during the week.
  Interventions: Other: Sensor Augmented Pump Therapy

INTERVENTIONS:
Device: DiAs — DiAs is the central component of our system. It is a standard cell phone running on an Android operating system. The cell phone has been changed to prevent from (1) using it as a phone or browser, (2) changing the volume (3) accidentally shutting it off. The cell phone runs an algorithm and is connected to work with the insulin pump and continuous glucose monitor to help keep the blood sugar in a desired range and help avoid hypoglycemia during the night.
  Arms: USS Virginia Closed Loop Control
Other: Sensor Augmented Pump Therapy — Insulin pump plus CGM.
  Other Names: SAP
  Arms: Sensor Augmented Pump Therapy

SUMMARY:
The purpose of this study is to use the USS Virginia Closed-Loop system for overnight insulin delivery in adults with Type 1 Diabetes (T1DM) in an outpatient setting to evaluate the system's ability to significantly improve blood glucose levels. This protocol will test the feasibility of "bedside" closed-loop control - an approach comprised of standard sensor-augmented pump therapy during the day using off-the-shelf devices and overnight closed-loop control using experimental devices in an outpatient setting. The rationale for this study is as follows: we anticipate that closed-loop control may ultimately be adopted by patients with T1DM in a selective manner. Patient may choose to start using these systems for overnight control only, e.g. to alleviate the well documented fear of hypoglycemia while asleep. To test this paradigm of "bedside" closed-loop control, subjects will be studied with continuous glucose monitoring (CGM)-augmented usual pump therapy during the day followed by overnight use of USS Virginia Closed Loop Control.

DETAILED DESCRIPTION:
The subject will participate in both the Experimental and the Control Admissions. The order of the two admissions will be randomized. During the Control Admission at home, the subject will use the study insulin pump along with a continuous glucose monitor receiver. During the Experimental Admission, the subject will be the research house/hotel where the subject will be in control of the DiAs. Participation in this study will require 5 study visits over 11-14 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis, based on investigator assessment, of type 1 diabetes for at least one year and using insulin for at least 1 year and an insulin pump for at least 6 months

   - Criteria for documented hyperglycemia (at least 1 must be met): i. Fasting glucose ≥126 mg/dL ii. Two-hour Oral Glucose Tolerance Test (OGTT) glucose ≥200 mg/dL iii. HbA1c ≥6.5% documented iv. Random glucose ≥200 mg/dL with symptoms v. No data at diagnosis is available but the participant has a convincing history of hyperglycemia consistent with diabetes.

   - Criteria for requiring insulin at diagnosis (1 must be met): i. Participant required insulin at diagnosis and continually thereafter ii. Participant did not start insulin at diagnosis but upon investigator review likely needed insulin (significant hyperglycemia that did not respond to oral agents) and did require insulin eventually and used continually iii. Participant did not start insulin at diagnosis but continued to be hyperglycemic, had positive islet cell antibodies - consistent with latent autoimmune diabetes in adults (LADA) and did require insulin eventually and used continually
2. Age ≥21 to <65 years
3. HbA1c <10.0%
4. For females, not currently known to be pregnant If female and sexually active, must agree to use a form of contraception to prevent pregnancy while a participant in the study. A negative urine pregnancy test will be required for all premenopausal women who are not surgically sterile. Subjects who become pregnant will be discontinued from the study.
5. Demonstration of proper mental status and cognition for the study
6. Currently using insulin-to-carbohydrate ratio to calculate meal bolus sizes
7. Ability to access the Internet and upload CGM data via the DexCom company software during the data collection period.
8. Willingness to remain within approximately 30 miles radius of study site during the day time hours of Visit 4.
9. An understanding of and willingness to follow the protocol and sign the informed consent

Additional Inclusion Criteria for UVA subjects only who participate in the 5 days at-home portion

* Availability of a significant other or family member committed to participating in all training activities, knowledgeable at all times of the participant's location, and being present and available to provide assistance when system is being used at night
* Commitment to maintaining uninterrupted availability via cell phone and avoiding any overnight travel for the duration of the period of time using the closed-loop system at home.
* Access to internet and cell phone service at home

Exclusion Criteria:

1. Admission for diabetic ketoacidosis in the 12 months prior to enrollment
2. Severe hypoglycemia resulting in seizure or loss of consciousness in the 12 months prior to enrollment
3. History of a seizure disorder (except hypoglycemic seizure), unless written clearance is received from a neurologist
4. Coronary artery disease or heart failure, unless written clearance is received from a cardiologist
5. Cystic fibrosis
6. A known medical condition that in the judgment of the investigator might interfere with the completion of the protocol such as the following examples:

   * Inpatient psychiatric treatment in the past 6 months
   * Presence of a known adrenal disorder
   * Abnormal liver function test results (Transaminase >2 times the upper limit of normal); testing required for subjects taking medications known to affect liver function or with diseases known to affect liver function
   * Abnormal renal function test results (calculated GFR <60 mL/min/1.73m2); testing required for subjects with diabetes duration of greater than 5 years post onset of puberty
   * Active gastroparesis
   * If on antihypertensive, thyroid, anti-depressant or lipid lowering medication, lack of stability on the medication for the past 2 months prior to enrollment in the study
   * Uncontrolled thyroid disease (TSH undetectable or >10 mlU/L); testing required within three months prior to admission for subjects with a goiter, positive antibodies, or who are on thyroid hormone replacement, and within one year otherwise
   * Abuse of alcohol or recreational drugs
   * Infectious process not anticipated to resolve prior to study procedures (e.g. meningitis, pneumonia, osteomyelitis).
   * Uncontrolled arterial hypertension (Resting diastolic blood pressure >90 mmHg and/or systolic blood pressure >160 mmHg).
   * Oral steroids
   * Uncontrolled microvascular complications such as current active proliferative diabetic retinopathy defined as proliferative retinopathy requiring treatment (e.g. laser therapy) in the past 12 months.
7. A recent injury to body or limb, muscular disorder, use of any medication, any carcinogenic disease, or other significant medical disorder if that injury, medication or disease in the judgment of the investigator will affect the completion of the protocol
8. Basal Rates <0.01 units/hour.
9. Current use of the following drugs and supplements:

   * Acetaminophen
   * Any medication being taken to lower blood glucose, such as Pramlintide, Metformin, glucagon-like peptide (GLP)-1 Analogs such as Liraglutide, and nutraceuticals intended to lower blood glucose
   * Beta blockers
   * Any other medication that the investigator believes is a contraindication to the subject's participation

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2014-06; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sue Brown, MD, Principal Investigator — University of Virginia; Carol Levy, MD, CDE, Principal Investigator — MOUNT SINAI HOSPITAL; Yogish C. Kudva, MBBS, MD, Principal Investigator — Mayo Clinic; Claudio Cobelli, PhD, Principal Investigator — University of Padova
Locations (4):
- United States (3):
  - Mayo Clinic, Rochester, Minnesota
  - Mount Sinai Hospital, New York, New York
  - University of Virginia Center for Diabetes Technology, Charlottesville, Virginia
- University of Padova, Padua, Italy

IPD SHARING:
Plan to Share IPD: Undecided
Undetermined

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: These results for 40 participants who completed the trial represent the combined results from participants at UVA, Mt. Sinai and Mayo Clinic (NCT02131766) combined with participants at University of Padua in Italy (NCT02008188).
Groups:
- USS Virginia Closed Loop Control and SAP: The subject will be admitted to the research house/hotel and will be discharged after 5 nights. The subject will be trained on DiAs and on how to respond to the system's alerts. The DiAs will be initiated by 11:00 PM and will be discontinued before breakfast. The staff will be monitoring the subject remotely. The subject will need to remain within a 30 miles of the research house/hotel during the day and return by 6:00 PM.
  A limited number of UVA and UPadova subjects will be asked to wear the DiAs at home for 5 days at the conclusion of research house admission.
  DiAs: DiAs is the central component of our system. It is a standard cell phone running on an Android operating system. The cell phone has been changed to prevent from (1) using it as a phone or browser, (2) changing the volume (3) accidentally shutting it off. The cell phone runs an algorithm and is connected to work with the insulin pump and continuous glucose monitor to help keep the blood sugar in a desired range and
Period: Overall Study
Arm/Group | USS Virginia Closed Loop Control and SAP
Started | 44
Completed | 40
Not Completed | 4
Not completed — Withdrawal by Subject | 4

BASELINE CHARACTERISTICS:
Groups:
- USS Virginia Closed Loop Control vs SAP: This is a cross-over trial in which each subject participates in two phases: USS Virginia Closed Loop Control (CLC) and Sensor Augmented Pump Therapy (SAP) and is randomized to order.
  During CLC: The subject will be admitted to the research house/hotel and will be discharged after 5 nights. The DiAs (CLC controller) will be initiated by 11:00 PM and will be discontinued before breakfast.
  During SAP: The subject will wear the continuous glucose monitor with the study insulin pump for a full 7 day period (approximately 7 consecutive 24 hour periods). The subject will follow their usual regimen.
  A limited number of UVA and UPadova subjects will be asked to wear the DiAs at home for 5 days at the conclusion of research house admission.
Arm/Group | USS Virginia Closed Loop Control vs SAP
Number analyzed (Participants) | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.5 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 18
Region of Enrollment [Number; unit: participants]
  United States | 28
  Italy | 12

OUTCOME MEASURES:

1. Primary Outcome: USS Virginia Time Within Target
Description: Assess the effect size of USS Virginia in increasing time within target (70-180 mg/dL) over a 24-hour period with closed-loop control overnight (23:00 to 07:00) as compared to sensor-augmented pump alone.
Time Frame: 40 hours
Population: Cross-over trial with same subjects participating in both arms for a total of 40 subjects.
Measure: Mean (Standard Deviation); unit: percentage of time spent in range
Groups:
- USS Virginia Closed Loop Control: The subject will be admitted to the research house/hotel and will be discharged after 5 nights. The subject will be trained on DiAs and on how to respond to the system's alerts. The DiAs will be initiated by 11:00 PM and will be discontinued before breakfast. The staff will be monitoring the subject remotely. The subject will need to remain within a 30 miles of the research house/hotel during the day and return by 6:00 PM.
  A limited number of UVA and UPadova subjects will be asked to wear the DiAs at home for 5 days at the conclusion of research house admission.
  DiAs: DiAs is the central component of our system. It is a standard cell phone running on an Android operating system. The cell phone has been changed to prevent from (1) using it as a phone or browser, (2) changing the volume (3) accidentally shutting it off. The cell phone runs an algorithm and is connected to work with the insulin pump and continuous glucose monitor to help keep the blood sugar in a desired range and
Arm/Group | USS Virginia Closed Loop Control | Sensor Augmented Pump Therapy
Number analyzed (Participants) | 40 | 40
percentage of time spent in range | 78.3 (10.2) | 71.4 (11.6)

2. Secondary Outcome: Overnight Target Range
Description: Assess time spent within target range of 80-140 mg/dl overnight with USS Virginia Closed Loop compared to sensor-augmented pump therapy alone
Time Frame: 40 hours
Population: Cross-over trial for a total of 40 participants
Measure: Mean (Standard Deviation); unit: percentage of time overnight
Groups:
- USS Virginia Closed Loop Control: The subject will be admitted to the research house/hotel and will be discharged after 5 nights. The subject will be trained on DiAs (CLC controller) and on how to respond to the system's alerts. The DiAs will be initiated by 11:00 PM and will be discontinued before breakfast.
  A limited number of UVA and UPadova subjects will be asked to wear the DiAs at home for 5 days at the conclusion of research house admission.
- Sensor Augmented Pump Therapy: The subject will wear the continuous glucose monitor with the study insulin pump for a full 7 day period (approximately 7 consecutive 24 hour periods).
  Sensor Augmented Pump Therapy: Insulin pump plus CGM.
Arm/Group | USS Virginia Closed Loop Control | Sensor Augmented Pump Therapy
Number analyzed (Participants) | 40 | 40
percentage of time overnight | 61.1 (20.6) | 39.6 (18.3)

3. Secondary Outcome: Decreased Overnight Hypoglycemia
Description: Assess the effect of USS Virginia Closed Loop System to decrease hypoglycemia overnight compared to sensor-augmented pump therapy alone
Time Frame: 40 hours
Population: Cross-over trial with a total of 40 participants
Measure: Mean (Standard Deviation); unit: percentage of time overnight
Arm/Group | USS Virginia Closed Loop Control | Sensor Augmented Pump Therapy
Number analyzed (Participants) | 40 | 40
percentage of time overnight | 0.9 (1.5) | 3.2 (3.4)

4. Secondary Outcome: Morning Glucose Levels
Description: Assess the distribution of wake-up glucose levels at 07:00 achieved by USS Virginia Closed Loop vs. to sensor-augmented pump therapy alone;
Time Frame: 40 hours
Population: Cross-over trial with a total of 40 participants
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | USS Virginia Closed Loop Control | Sensor Augmented Pump Therapy
Number analyzed (Participants) | 40 | 40
mg/dL | 123.7 (17.8) | 145.3 (31.0)

ADVERSE EVENTS:
Time Frame: Approximately 2-3 weeks.
Groups:
- USS Virginia Closed Loop Control and SAP: Combined Group in Cross-Over Trial that had CLC and SAP.
Arm/Group | USS Virginia Closed Loop Control and SAP
Serious Adverse Events (participants affected / at risk) | 0/40
Other Adverse Events (participants affected / at risk) | 1/40
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | USS Virginia Closed Loop Control and SAP (N=40)
Otitis media (Ear and labyrinth disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No